CLINICAL TRIAL: NCT06866301
Title: DiANa Project: Uncovering the Relationship Between MircroRNA Expression, Gut Microbiota and Prognosis in Patients with Anorexia Nervosa.
Brief Title: Active Lifestyle Intervention in Anorexia Nervosa: a Comprehensive Study
Acronym: DiANa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SV-PA-21-AYUD/2021/58376
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; microRNA; Gut Microbiota; Exercise; Physical Fitness; Mental Health; Body Composition
MeSH Terms: conditions — Anorexia Nervosa; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AN-Intervention (Experimental): Patient enrolled in the exercise intervention group
  Interventions: Behavioral: Progressive Resistance Exercise
- AN-Control (No Intervention): Patient enrolled in the non-exercise group
- H-Control (No Intervention): Healthy controls in the non-exercise group

INTERVENTIONS:
Behavioral: Progressive Resistance Exercise — The exercise program will have a duration of 10 weeks. It will be divided in two phases: conditioning phase and training phase. During the conditioning phase (2-3 weeks), participants will learn exercise techniques, work on their interoceptive awareness and perform same exercises at a lower intensity to prepare the muscles for the next phase. In the training phase, the intensity will be moderate starting at approximately 60% of capacity, with a frequency of three days per week and continuous adjustment (progression) based on the participant's improvements. Each session will include a warm-up and cool-down of approximately 10 minutes. The central part of the session will be in the form of a circuit and will include 6 large muscle group exercises using a combination of machine exercises following the PPL (push, pull and legs) model and 3 core strengthening exercises.
  Arms: AN-Intervention

SUMMARY:
The goal of this study is to perform a comprehensive analysis of varied health markers and analyze the impact of lifestyle interventions on the prognosis of anorexia nervosa (AN) patients. In addition, this study aims to determine if biomarker analysis can be used as clinical outcomes for disease prognosis long-term and support individualized treatment strategies in female patients with AN during the post-hospitalization phase.

The main questions it aims to answer are:

* What are the miRs and microbiota profiles associated with AN, and how are they linked to other clinical markers?
* How does a lifestyle intervention (exercise with nutritional support) affect biomarkers and clinical markers during the first three months after hospitalization?
* What are the dynamics and associations of biomarkers, including gut microbiota, and how do they relate to critical events during the six months after hospitalization?
* What is the perceived effect of participating in a healthy lifestyle program for patients, families, and professionals involved in the care of these patients?

Participants will:

* Undergo analysis of biomarkers and gut microbiota associated with AN.
* Participate in a lifestyle intervention program involving exercise during the first three months post-hospitalization.
* Provide samples for biomarker and gut microbiota mapping over a six-month period.
* Share feedback on their perceived experience in the lifestyle program through interviews or surveys.

Researchers will compare biomarker and gut microbiota and the effects of the intervention to determine if a lifestyle exercise intervention can lead to better outcomes, and analyze its potential to individualized care strategies.

ELIGIBILITY:
Inclusion Criteria:

A) Patients:

* Patients with a diagnosis of AN (any subtype)
* BMI >14kg/m2
* Under treatment at the Regional Eating Disorders Unit at the Area IV and V of the Principality of Asturias
* After acute treatment (total or partial hospitalization or other acute treatment regime following the recommendation of the medical team)

B) Healthy Controls:

- Meet the physical activity recommendations of the World Health Organization for the age group and sex.

Exclusion Criteria:

A) Patients:

* Contraindications to perform the evaluations proposed in this project
* Unmanaged dysfunctional or compulsive exercise
* Other criteria that, in the opinion of the medical team, prioritize the patient's health (i.e., psychological instability, substance abuse) .

B) Healthy Controls:

* Suffer from metabolic, pulmonary or cardiovascular disease
* Suffer from serious organic disease
* Taking prescribed medications while participating in the project
* Have contraindications to perform the proposed assessments or intervention.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of microRNA profile from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  microRNAs are epigenetic markers that are sensitive to lifestyle interventions. A possible change is an improved profile after exercise intervention. microRNAs are measured in reads per million
Change of gut microbiota profile from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Gut microbiota is a group of bacteria that are sensitive to lifestyle interventions, stress and other environmental factors. A possible change is an improved profile after exercise intervention. Microbiota is measured in reads per million
Change of Eating Disorders Examination Questionnaire (EDE-Q) scores from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  The EDE-Q provides a global score and four subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) derived from a 7-point Likert scale, where 0 indicates no symptoms or concerns and 6 indicates the most severe symptoms or concerns. Higher scores represent greater severity of eating disorder pathology
Change of muscle strength from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Muscle strength is a physical fitness marker that is sensitive to lifestyle interventions. A possible change is an improved muscle strength after exercise intervention. Strength is measured in kilograms, Newtons, Watts, velocity (meters/second) or time (seconds).
Change of muscle content from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Muscle content is a marker of health that is sensitive to lifestyle interventions and is measured with BioImpedance Analysis. A possible change is an improved muscle content after exercise intervention. Muscle content is measured in Kilograms or squared centimeters.

SECONDARY OUTCOMES:
Change of the anthropometric profile from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Anthropometric measurements server as a marker of body composition which are sensitive to lifestyle interventions. A possible change is an improved anthropometric profile after exercise intervention. Anthropometric variables are measured in kilograms (body weight), meters (height), centimeters (circumferences), millimeters (skinfolds).
Change of fat content from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Fat content is a health marker that is sensitive to lifestyle interventions. A possible change is an improved fat content after exercise intervention and is measured with BioImpedance Analysis. Fat content is measured in kilograms or millimeters.
Change of functional capacity from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Functional capacity is a marker that indicates the capacity of the body to supply oxygen and nutrients to the muscles for energy production. It is sensitive to lifestyle interventions. A possible change is an improved functional capacity after exercise intervention. Functional capacity is measured in milliliters per kilogram per minute, Liters per minute, meters per second, beats per minute, or time (minutes).
Change of Physical Activity Levels from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  Physical Activity Levels are markers of health and well-being sensitive to lifestyle interventions. A possible change is an improved physical activity level profile after exercise intervention. Physical activity levels are measured in minutes/day, kcals, counts or % of time during the day/week.
Change of Beck Depression Inventory 2 (BDI-2) from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  The Beck Depression Inventory-2 (BDI-2) is a self-report questionnaire designed to assess the severity of depressive symptoms. Each item is rated on a 4-point scale ranging from 0 to 3, where 0 indicates no symptom severity and 3 indicates the most severe level of the symptom. The total score ranges from 0 to 63, with higher scores indicating greater severity of depressive symptoms.
Change of Brief Symptom Inventory (BSI) scores from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  The Brief Symptom Inventory (BSI) is a self-report questionnaire designed to assess distress across three symptom dimensions (depression, anxiety, and somatization) and a global severity index. Higher scores reflect greater levels of distress or severity of symptoms.
Change of The Short Form-36 Health Survey (SF-36) scores from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  The Short Form-36 Health Survey (SF-36) is a self-report questionnaire designed to measure health-related quality of life across eight domains (Physical Functioning, Role Limitations due to Physical Health, Role Limitations due to Emotional Problems, Energy/Fatigue, Emotional Well-being, Social Functioning, Pain, and General Health). Scores for each domain, as well as a physical and mental component summary score, are derived on a scale from 0 to 100, where 0 indicates the worst possible health or functioning and 100 indicates the best possible health or functioning. Higher scores reflect better health and quality of life.

OTHER OUTCOMES:
Change of Exercise Dependence Scale-Revised (EDS-R) scores from baseline to week 12 and week 24 | Baseline, week 12 and week 24
  The Exercise Dependence Scale-Revised (EDS-R) is a self-report questionnaire used to assess symptoms of exercise dependence through seven subscales (Tolerance, Withdrawal, Continuance, Lack of Control, Reduction in Other Activities, Time, and Intention Effects). Rated on a 6-point Likert scale (1 indicates "Never", 6 indicates "Always"), higher scores indicate greater severity of exercise dependence symptoms.
Perceptions related to exercise resulted from the intervention after 24 weeks | After 24 weeks
  Perceptions of patients related to exercise are sensitive to lifestyle and educational interventions and are measured through guided interviews. A possible finding is an improved perception after exercise intervention. Interviews are analyzed throughout qualitative methods by categorizing common themes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of the data collected in this clinical trial, which involves individuals with eating disorders, including minors and young adults, we have decided not to share individual participant data (IPD). Eating disorders are highly stigmatized conditions, and although the data do not contain personally identifiable and health-related information, the population in the area is reduced so we want to prevent potential privacy risks, even with de-identification efforts. Additionally, the inclusion of underage participants necessitates strict adherence to ethical and legal protections regarding their confidentiality. Ensuring the privacy and well-being of this vulnerable population is our utmost priority, aligning with ethical guidelines and data protection regulations.